CLINICAL TRIAL: NCT01172756
Title: Acute Hemodynamic Effects of Riociguat (BAY63-2521) in Patients With Pulmonary Hypertension Associated With Diastolic Heart Failure: A Randomized, Double-blind, Placebo-controlled, Single-dose Study in Three Ascending Dose Cohorts
Brief Title: A Study to Test the Effects of Riociguat in Patients With Pulmonary Hypertension Associated With Left Ventricular Diastolic Dysfunction
Acronym: DILATE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was only stopped after the statistical power of the study was reached and the study objectives could be met despite the premature discontinuation.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14554; 2010-018436-41 (EudraCT Number)
Record Dates: First submitted 2010-07-19; First posted 2010-07-30 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Hypertension, Pulmonary; Ventricular Dysfunction, Left
Keywords: Pulmonary Hypertension; Left ventricular dysfunction
MeSH Terms: conditions — Hypertension, Pulmonary; Ventricular Dysfunction, Left | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Riociguat (BAY63-2521)
- Arm 2 (Experimental)
  Interventions: Drug: Riociguat (BAY63-2521)
- Arm 3 (Experimental)
  Interventions: Drug: Riociguat (BAY63-2521)
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riociguat (BAY63-2521) — 0.5 mg single oral dose
  Arms: Arm 1
Drug: Riociguat (BAY63-2521) — 1 mg single oral dose
  Arms: Arm 2
Drug: Riociguat (BAY63-2521) — 2 mg single oral dose
  Arms: Arm 3
Drug: Placebo — single oral dose
  Arms: Arm 4

SUMMARY:
The aim of this study is to assess whether single oral doses of Riociguat safely improve the cardiovascular function in patients with pulmonary hypertension associated with left ventricular diastolic dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with symptomatic pulmonary hypertension due to left ventricular diastolic dysfunction

Exclusion Criteria:

* Types of pulmonary hypertension other than group 2.2 of Dana Point Classification

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pulmonary artery mean pressure at rest | Peak change from baseline within 6 hours after a single dose of study drug

SECONDARY OUTCOMES:
Adverse event collection | until 30 days after study drug treatment
Plasma concentrations to obtain pharmacokinetic profile of Riociguat | Within 24 hours after study drug treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Austria (4):
  - Graz, Styria
  - Linz, Upper Austria
  - Vienna, Vienna
  - Salzburg
- Prague, Czechia
- Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Bonderman D, Pretsch I, Steringer-Mascherbauer R, Jansa P, Rosenkranz S, Tufaro C, Bojic A, Lam CSP, Frey R, Ochan Kilama M, Unger S, Roessig L, Lang IM. Acute hemodynamic effects of riociguat in patients with pulmonary hypertension associated with diastolic heart failure (DILATE-1): a randomized, double-blind, placebo-controlled, single-dose study. Chest. 2014 Nov;146(5):1274-1285. doi: 10.1378/chest.14-0106. PMID 24991733
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu